CLINICAL TRIAL: NCT00053183
Title: Phase I Brachytherapy Dose Escalation Using The GliaSite RTS In Newly Diagnosed Glioblastoma Multiforme In Conjunction With External Beam Radiation Therapy
Brief Title: Surgery Followed by Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000269300; NABTT-2105; JHOC-NABTT-2105
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2004-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Brachytherapy; Radiotherapy

INTERVENTIONS:
Procedure: conventional surgery
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. External-beam radiation therapy uses high-energy x-rays to kill tumor cells. Combining internal radiation with external-beam radiation therapy may kill any remaining tumor cells following surgery.

PURPOSE: Phase I trial to study the effectiveness of combining internal radiation therapy with external-beam radiation therapy in treating patients who have undergone surgery for glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of brachytherapy administered via GliaSite RTS™ applicator followed by external beam radiotherapy in patients with newly diagnosed glioblastoma multiforme.
* Determine the acute and chronic toxicity of brachytherapy administered via GliaSite RTS™ in these patients.
* Determine the survival rate of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of brachytherapy.

Patients undergo craniotomy for histologic confirmation of glioblastoma multiforme, surgical resection, and placement of a GliaSite RTS™ applicator that includes Iotrex™.

Beginning 3-21 days after surgery, patients undergo brachytherapy via the GliaSite RTS™ applicator. Within 30 days of brachytherapy (no more than 60 days after resection) patients undergo external beam radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 5-10 patients receive escalating doses of brachytherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 5 or 3 of 10 patients experience dose-limiting toxicity.

Patients are followed at 21-35 days, every 2 months for 1 year, and then for survival.

PROJECTED ACCRUAL: A total of 15-100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically suspected supratentorial grade IV glioblastoma multiforme
* Candidate for maximal surgical resection of tumor mass

  * Expected residual enhancing tumor must be within the expected brachytherapy treatment volume
  * Resection must not be expected to result in a new permanent neurologic deficit
* No clearly multi-focal disease (2 or more separate foci of contrast-enhancing tumor not all within the expected brachytherapy prescription volume by MRI)
* No enhancing tumor greater than 1 cm beyond the midline by MRI
* No grossly or radiographically apparent leptomeningeal spread and/or ventricular invasion outside the anticipated radiation treatment volume
* No marked edema by MRI with significant shift that is not anticipated to be corrected by resection

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine no greater than 1.7 mg/dL
* BUN no greater than 2 times upper limit of normal

Cardiovascular

* No uncontrolled hypertension
* No unstable angina pectoris
* No uncontrolled cardiac dysrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Mini mental state exam score at least 15
* No other concurrent medical illness that would preclude study participation
* No concurrent serious infection
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No immunotherapy prior to, during, or within 90 days after brachytherapy
* No biologic therapy with any of the following prior to, during, or within 90 days after brachytherapy :

  * Immunotoxins
  * Immunoconjugates
  * Antiangiogenesis compounds
  * Peptide receptor antagonists
  * Interferons
  * Interleukins
  * Tumor-infiltrating lymphocytes
  * Lymphokine-activated killer cells
  * Gene therapy
  * Antisense agents

Chemotherapy

* No chemotherapy or polifeprosan 20 with carmustine implant (Gliadel wafers) prior to, during, or within 90 days after brachytherapy

Endocrine therapy

* No hormonal therapy prior to, during, or within 90 days after brachytherapy
* Concurrent corticosteroids to improve quality of life allowed

Radiotherapy

* No other radiotherapy prior to, during, or within 90 days after brachytherapy

Surgery

* See Disease Characteristics
* No radiosurgery prior to, during, or within 90 days after brachytherapy

Other

* No other investigational agents directed at the brain tumor prior to, during, or within 90 days after brachytherapy
* Concurrent noncytotoxic therapy to improve quality of life allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Volker W. Stieber, MD, Study Chair — Wake Forest University Health Sciences
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas